CLINICAL TRIAL: NCT01107327
Title: FDG PET in Cancer Associated Venothromboembolism
Brief Title: Fluorodeoxyglucose (FDG)-Positron Emission Tomography (PET) in Cancer Associated Venothromboembolism
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HCI18327; R01CA121003-01 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-04-20 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Venothromboembolism
Keywords: cancer
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: FDG-PET/CT — The study is focused on two goals, both of which use a new imaging test called PET/CT. PET/CT combines a special radioactive scan with a CT scan. PET/CT is most commonly used in medical practice to evaluate cancer. Abnormal areas such as cancer "light up" on the PET/CT scan. However, many doctors, including us, have noticed that PET/CT also "lights up" in areas of blood clot formation as well. In this study, PET/CT will be used to evaluate the two goals of this project.
  Other Names: PET scan,; PET/CT scan; FDG-PET/CT scan; FDG-PET

SUMMARY:
Venothromboembolic disease (VTE), which includes deep venous thrombosis (DVT) and pulmonary embolism (PE), is a severe health problem, effecting 1.5/1000 per year in the general population. In patients over 60 years of age, the incidence is 1/100 per year. Of the two million Americans per year who will develop VTE, one third will develop pulmonary embolism (PE). VTE is usually diagnosed by Doppler ultrasound or contrast venography when present in the extremities, VQ scan or pulmonary angiography when PE is present. However, there are many instances when the diagnosis of VTE by conventional modalities is limited. These include obesity, recent trauma or surgery, the presence of a mass, the presence of clot around central lines, and clot occurring in the abdomen and pelvis. Furthermore, the differentiation between new and old clot has evaded all diagnostic imaging modalities, and no existing modality allows for an accurate delineation of all sites of thrombus within the body. New approaches to the diagnostic imaging of VTE in complicated cases are needed. The first hypothesis of this project is that FDG PET/CT can be used to accurately diagnose the presence and extent of acute VTE, and that it will distinguish new clot from old.

Approximately 20-25% of all new cases of venous thromboembolism occur in known cancer patients. The risk of VTE is 4-6 fold greater in patients with cancer as those without (8-12% vs. 2%, respectively, lifetime risk). In many cases, the development of VTE occurs as the first clinical sign of the cancer, even before it is diagnosed. Among patients presenting with acute VTE have no obvious cause (defined as "idiopathic" or "unprovoked", as opposed to "secondary" VTE), the literature reports that up to 20% (range of reported incidence 7-20%) may ultimately prove to have cancer, depending on the series and whether the thrombosis is unifocal or multifocal. Despite the substantial prevalence of occult cancer in patients presenting with idiopathic VTE, there are no current recommendations that these patients be screened for the presence of cancer. The second hypothesis of the project is that FDG PET/CT can accurately be used to screen for the presence of cancer in patients with unprovoked (idiopathic) acute VTE.

Objectives:

There are two specific objectives to test the hypotheses associated with this project:

1. To establish the sensitivity of FDG PET/CT in the diagnosis of acute VTE.
2. To perform a pilot project to aid in the design of a larger trial to define the incidence of occult cancer in patients rigorously selected for idiopathic (unprovoked) VTE, and to investigate the value of FDG PET in the early detection of occult cancer in this population.

DETAILED DESCRIPTION:
Study AIM #1 To establish the sensitivity of FDG PET/CT in the diagnosis of acute VTE.

Rationale: We believe that FDG PET/CT can be used to accurately diagnose the presence, extent, and acuity of VTE. It is unrealistic to assume that FDG-PET could or should become the primary imaging modality for evaluating VTE. The cost, compared to Doppler ultrasound, would be prohibitive, and would involve unnecessary radiation of the patient. We intend to establish the value of FDG PET, instead, as an alternative modality for the diagnosis of VTE. Clinical situations where this might prove useful include: 1) the presence of old clot, when the distinction between new and old may be important; 2) evaluation of abdominal, pelvic and thoracic thrombus, where Doppler is difficult-to-impossible because of patient obesity; 3) Complicated anatomy due to the presence of tumor or post-therapeutic changes.

The sensitivity of FDG PET/CT will be established in patients with acute VTE. The accuracy with which sites of abnormal FDG uptake can be related, spatially, to vascular structures will be critical to the success of this study. There is little doubt that this can better be accomplished with PET/CT than with PET alone. PET/CT will be used for all of these studies. Patients with documented acute VTE, will be enrolled. To determine the utility of FDG PET/CT in distinguishing acute from subacute or chronic clot, and to establish the extent of acute clot, the initial whole body PET/CT scan must be performed within 2 weeks of onset of symptoms of DVT, and subsequent limited region PET/CT scans will be performed at 2-3 weeks and at 6 weeks following the initial PET/CT scan. Whenever possible, subjects will be recruited who have unprovoked VTE because the potential benefit to the patient for participating in this study will be greatest for these patients are at a higher risk for harboring an underlying occult malignancy. However, patients with both provoked and unprovoked VTE will be eligible for enrollment under this specific aim.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria will include documented acute DVT (+/-PE) by Doppler ultrasound or contrast venography.
2. Subjects will be eligible either with provoked or unprovoked DVT.
3. To meet the inclusion criteria, patients must be enrolled and the initial PET/CT scan performed within 2 weeks of initial onset of symptoms of VTE.

Exclusion Criteria:

1. Subjects less than 18 years of age,
2. Those who are unable to understand and provide signature informed consent
3. Pregnant subjects. Any female of childbearing age who has a uterus and functional ovaries will undergo a serum pregnancy test prior to inclusion. 4. Subjects with calf-only blood clot will be excluded, due to the fact that these cases are often complicated by venous stasis disease, post-phlebitic syndrome, and the presence of both acute and chronic clot, which may compromise interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be eligible either with provoked or unprovoked DVT.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of FDG PET/CT scanning to diagnose presence, extent, and acuity of Ventothromboembolism diagnosis. | April 2012
  We believe that FDG PET/CT can be used to accurately diagnose the presence, extent, and acuity of VTE. We intend to establish the value of FDG PET, instead, as an alternative modality for the diagnosis of VTE. Clinical situations where this might prove useful include: 1) the presence of old clot, when the distinction between new and old may be important; 2) evaluation of abdominal, pelvic and thoracic thrombus, where Doppler is difficult-to-impossible because of patient obesity; 3) Complicated anatomy due to the presence of tumor or post-therapeutic changes.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Morton, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Rondina MT, Lam UT, Pendleton RC, Kraiss LW, Wanner N, Zimmerman GA, Hoffman JM, Hanrahan C, Boucher K, Christian PE, Butterfield RI, Morton KA. (18)F-FDG PET in the evaluation of acuity of deep vein thrombosis. Clin Nucl Med. 2012 Dec;37(12):1139-45. doi: 10.1097/RLU.0b013e3182638934. PMID 23154470